CLINICAL TRIAL: NCT00004779
Title: Phase I Pilot Study of Ad5-CB-CFTR, an Adenovirus Vector Containing the Cystic Fibrosis Transmembrane Conductance Regulator Gene, in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of North Carolina (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11829; UNCCH-921
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

INTERVENTIONS:
Genetic: Ad5-CB-CFTR

SUMMARY:
OBJECTIVES: I. Assess the safety and efficacy of gene transfer into the nasal epithelium using Ad5-CB-CFTR, an E1-deleted adenovirus vector containing the cystic fibrosis transmembrane conductance regulator gene, in patients with cystic fibrosis (CF).

II. Determine whether ion transport abnormalities in CF airway cells can be corrected.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Groups of 3 patients receive 1 of 4 doses of Ad5-CB-CFTR, a recombinant E1-deleted adenovirus serotype 5 vector containing the cystic fibrosis transmembrane conductance regulator gene. Ad5-CB-CFTR is administered to 1 nasal cavity and the vehicle alone is administered to the opposite nasal cavity as the control.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Cystic fibrosis No mild genetic mutations, i.e., normal nasal chloride ion permeability At least 2 weeks since decrease in pulmonary function --Prior/Concurrent Therapy-- At least 3 months since systemic cortisone At least 1 month since other therapeutic research study, e.g., DNAse --Patient Characteristics-- Other: Adequate endocrine, liver, kidney, and cardiac function Adenovirus antibody seropositive No pregnant or nursing women Negative pregnancy test required of fertile women Adequate contraception required of fertile patients

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 1993-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Knowles, Study Chair — University of North Carolina